CLINICAL TRIAL: NCT03944473
Title: Accessor Blinded Randomized Controlled Study Evaluating the Efficacy and Safety of Sugammadex in High-Risk Ambulatory Surgeries
Brief Title: Efficacy and Safety of Sugammadex in High-Risk Ambulatory Surgeries
Acronym: Sugammadex
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped before IRB approval
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Curtis Choice, Director, Ambulatory Anesthesia Division, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019-10223
Record Dates: First submitted 2019-04-30; First posted 2019-05-09 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Ambulatory Difficulty
Keywords: high risk; chronic health condition; laparoscopic surgery
MeSH Terms: conditions — Mobility Limitation | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: On the day of surgery, an envelope containing the randomization code will be given to an anesthesiology physician or nurse anesthetist responsible for the clinical care of the study patient. Patients will be randomly allocated to receive neostigmine or sugammadex using a 1:1 allocation ratio. Patients will be stratified based on their ASA physical score. A research associate who is not directly involved with the study procedures will maintain the randomization codes. All others will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- neostigmine (Active Comparator): Neostigmine is the acetylcholinesterase inhibitor most commonly used in pharmacologically reversing the effects of neuromuscular blockers [8]. Reversal of NMB is facilitated by increasing acetylcholine levels at nicotinic skeletal muscle-binding sites.
  Interventions: Drug: Neostigmine
- sugammadex (Experimental): Sugammadex is a modified gamma-cyclodextrin, the first of a new class of drugs called selective relaxant binding agents, with an unusually high affinity for rocuronium. This medication offers an alternate mechanism of action to antagonize the effects of steroidal neuromuscular blockade agents.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Patients undergoing laparoscopic ambulatory surgery randomized into Sugammadex group will receive a dose of Sugammadex as their reversal agent
  Arms: sugammadex
Drug: Neostigmine — Patients undergoing laparoscopic ambulatory surgery randomized into Neostigmine group will receive a dose of Neostigmine as their reversal agent
  Arms: neostigmine

SUMMARY:
In this randomized controlled study, the investigators hypothesize that sugammadex is superior to neostigmine in higher risk patients undergoing laparoscopic outpatient surgery in an urban, stand-alone ambulatory surgery center.

The primary objective of this study is to evaluate the "fit to discharge time in the PACU." The secondary objectives are PACU adverse events, use of additional medications in the PACU, 0-30 day ED or inpatient admissions for a pulmonary diagnosis and patient satisfaction at discharge.

DETAILED DESCRIPTION:
There is limited published data in the use of sugammadex for high-risk patient populations, such as those undergoing laparoscopic procedures in standalone outpatient surgery facilities. About 90% of the ambulatory surgical patient population at this institution is non-caucasian with the majority of the higher-risk patients having obesity and one or more additional chronic health conditions. In this randomized controlled study, the investigators hypothesize that sugammadex is superior to neostigmine in higher risk patients undergoing laparoscopic outpatient surgery in an urban, stand-alone ambulatory surgery center.

The primary objective of this study is to evaluate the "fit to discharge time in the PACU." The secondary objectives are PACU adverse events, use of additional medications in the PACU, 0-30 day ED or inpatient admissions for a pulmonary diagnosis and patient satisfaction at discharge.

In this double-blinded randomized controlled study, the study team is evaluating the efficacy and safety of sugammadex in patients undergoing ambulatory surgical procedures. Currently, both neostigmine and sugammadex are standard of care in this institution. Other than the emergent need for NMB reversal, practice preference and individual indications dictate the selection of reversal medication.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical score II and III
* Scheduled for a laparoscopic ambulatory surgery
* 21-60 years of age
* Able to understand and sign informed consent

Exclusion Criteria:

* Known allergy to neostigmine or sugammadex
* Active pulmonary diagnosis
* American Society of Anesthesia physical score 4 and above
* Known or suspected neuromuscular disease
* Documented renal or liver insufficiency (2 fold increase in the labs)
* Body Mass Index >40
* Any surgical case brought into the operating room after 4 PM (to avoid any provider bias related to discharging patients before closure of the ambulatory surgery center for the day)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-07-20 (Estimated)

PRIMARY OUTCOMES:
Aldrete Score | Up to 5 hours
  The Aldrete Score will determine transfer from phase 1 to phase 2 recovery. The following criterias will be scored from 0 to 2- activity level, respiration, blood pressure, consciousness, oxygen saturation. Patients who get a total score of 9 or more are considered ready for discharge from Post Anesthesia Care Unit
Post Anesthetic Discharge Scoring System | Up to 5 hours
  The Post Anesthetic Discharge Scoring System (PADSS) will be used to determine discharge to home readiness. Six criterias to score- vital signs, ambulation, nausea/vomiting, pain, bleeding and voiding. Each one is given a score from 0 to 2. Patients who get a total score of 9 or more are considered ready for discharge from Post Anesthesia Care Unit
Fit To PACU Discharge | Up to 5 hours
  Based on Post Anesthetic Discharge Scoring System (PADSS), the primary outcome measure will be calculated as the time from study medication administration to the time of "fit to discharge from Post Anesthesia Care Unit (PACU)."

SECONDARY OUTCOMES:
Rate of adverse events in PACU | Up to 5 hours
  The research associate will record the adverse events related to delay in discharge during stay in Post Anesthesia Care Unit (PACU)
use of additional medications in PACU | Up to 5 hours
  The research associate will record any medications used in the Post Anesthesia Care Unity (PACU).
Emergency Department or inpatient admissions within 30 days after discharge | 30 days after discharge
  One month ED visits and inpatient admissions for a pulmonary diagnosis will be collected from the medical records.
patient satisfaction | Up to 5 hours
  At the time of discharge from PACU when patients are fully recovered and conscious, a validated satisfaction survey will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Choice, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shnaider I, Chung F. Outcomes in day surgery. Curr Opin Anaesthesiol. 2006 Dec;19(6):622-9. doi: 10.1097/ACO.0b013e328010107e. PMID 17093366
- [Background] Hall MJ, Schwartzman A, Zhang J, Liu X. Ambulatory Surgery Data From Hospitals and Ambulatory Surgery Centers: United States, 2010. Natl Health Stat Report. 2017 Feb;(102):1-15. PMID 28256998
- [Background] Watkins AC, White PF. Fast-tracking after ambulatory surgery. J Perianesth Nurs. 2001 Dec;16(6):379-87. doi: 10.1053/jpan.2001.28887. PMID 11740779
- [Background] King M, Sujirattanawimol N, Danielson DR, Hall BA, Schroeder DR, Warner DO. Requirements for muscle relaxants during radical retropubic prostatectomy. Anesthesiology. 2000 Dec;93(6):1392-7. doi: 10.1097/00000542-200012000-00008. PMID 11149431
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Martinez-Ubieto J, Ortega-Lucea S, Pascual-Bellosta A, Arazo-Iglesias I, Gil-Bona J, Jimenez-Bernardo T, Munoz-Rodriguez L. Prospective study of residual neuromuscular block and postoperative respiratory complications in patients reversed with neostigmine versus sugammadex. Minerva Anestesiol. 2016 Jul;82(7):735-42. Epub 2015 Oct 16. PMID 26472231
- [Background] Fortier LP, McKeen D, Turner K, de Medicis E, Warriner B, Jones PM, Chaput A, Pouliot JF, Galarneau A. The RECITE Study: A Canadian Prospective, Multicenter Study of the Incidence and Severity of Residual Neuromuscular Blockade. Anesth Analg. 2015 Aug;121(2):366-72. doi: 10.1213/ANE.0000000000000757. PMID 25902322
- [Background] Brull SJ, Kopman AF. Current Status of Neuromuscular Reversal and Monitoring: Challenges and Opportunities. Anesthesiology. 2017 Jan;126(1):173-190. doi: 10.1097/ALN.0000000000001409. PMID 27820709
- [Background] Hyman EC, Brull SJ. Clarification: Current Status of Neuromuscular Reversal and Monitoring, Challenges and Opportunities. Anesthesiology. 2017 Oct;127(4):730. doi: 10.1097/ALN.0000000000001795. No abstract available. PMID 28926458
- [Background] Welliver M, Cheek D, Osterbrink J, McDonough J. Worldwide experience with sugammadex sodium: implications for the United States. AANA J. 2015 Apr;83(2):107-15. PMID 26016169
- [Background] Soto R, Jahr JS, Pavlin J, Sabo D, Philip BK, Egan TD, Rowe E, de Bie J, Woo T. Safety and Efficacy of Rocuronium With Sugammadex Reversal Versus Succinylcholine in Outpatient Surgery-A Multicenter, Randomized, Safety Assessor-Blinded Trial. Am J Ther. 2016 Nov/Dec;23(6):e1654-e1662. doi: 10.1097/MJT.0000000000000206. PMID 25768376
- [Background] Cho HC, Lee JH, Lee SC, Park SY, Rim JC, Choi SR. Use of sugammadex in lung cancer patients undergoing video-assisted thoracoscopic lobectomy. Korean J Anesthesiol. 2017 Aug;70(4):420-425. doi: 10.4097/kjae.2017.70.4.420. Epub 2017 Apr 21. PMID 28794837
- [Background] Sabo D, Jahr J, Pavlin J, Philip B, Shimode N, Rowe E, Woo T, Soto R. The increases in potassium concentrations are greater with succinylcholine than with rocuronium-sugammadex in outpatient surgery: a randomized, multicentre trial. Can J Anaesth. 2014 May;61(5):423-32. doi: 10.1007/s12630-014-0128-7. Epub 2014 Apr 8. PMID 24710957
- [Background] Kim YH. Sugammadex: watch out for new side effects. Korean J Anesthesiol. 2016 Oct;69(5):427-428. doi: 10.4097/kjae.2016.69.5.427. Epub 2016 Sep 8. No abstract available. PMID 27703621